CLINICAL TRIAL: NCT04387006
Title: Osteopathic Manipulative Treatment Induces Functional Connectivity Changes: a Randomized Manual Placebo-controlled Trial
Brief Title: Osteopathic Manipulative Treatment Induces Functional Connectivity Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Marco Tramontano, Head of Rehabilitation Services, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE/PROG625
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Osteopathic Manipulative Treatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopatic Manipulative Treatment (OMT) (Experimental)
  Interventions: Other: OMT
- Manual Placebo (MP) (Placebo Comparator)
  Interventions: Other: MP

INTERVENTIONS:
Other: OMT — OMT techniques were focused on correcting the dysfunctions found during the initial physical examination and included articular and myofascial techniques, balanced ligamentous tension, visceral manipulations and osteopathy in the cranial field
  Arms: Osteopatic Manipulative Treatment (OMT)
Other: MP — MP treatment was performed by the same osteopaths who performed OMT and was carried out in the same hospital setting. P treatment consisted of a passive touch without joint mobilization in a protocolled order. The osteopaths were standing next to the bed, they touched lumbar and dorsal spine of the subjects in prone position for 10 minutes, and then in supine position, they touched for 10 minutes the shoulders, the hips, then the neck, the sternum and the chest were touched for 5 minutes each. Another researcher on the placebo protocol specifically trained the osteopaths.
  Arms: Manual Placebo (MP)

SUMMARY:
Osteopathic Manipulative Treatment (OMT) is a whole-body intervention mainly focused on correcting the somatic dysfunctions present in different regions of the body. Osteopathic research to date has mostly been concerned with various clinical conditions such as musculoskeletal disorders and primary headache. The neurophysiological effects underlying clinical improvements are still under debate. Although models explaining the therapeutic effects of OMT include the potential for higher brain mechanism, OMT effects on functional brain connectivity is not fully understood and still lacking in healthy adults. Magnetic resonance imaging (MRI) research includes several different approaches to estimate cortical functions. Several of these approaches have demonstrated functional brain changes associated with OMT. Using Arterial Spin Labeling MRI, recently was demonstrated that the treatment of somatic dysfunctions induces cerebral perfusion changes in asymptomatic young participant. Thus, the aim of this study is to explore the neural correlates associated with OMT effect in terms of cerebral functional connectivity, as derived by complex network analysis of resting state fMRI data recorded in asymptomatic young volunteers with somatic dysfunctions

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 40 years
* suitability for MRI scanning

Exclusion Criteria:

* cognitive impairment, based on Mini Mental State Examination (MMSE) score ≤ 24 according to norms for the Italian population, and confirmed by a deeper clinical neuropsychological evaluation using the Mental Deterioration Battery and NINCDS-ADRDA criteria for dementia
* subjective complaints of memory difficulties or of any other cognitive deficit, interfering or not, with daily living activities;
* major medical illnesses, e.g., diabetes (not stabilized), obstructive pulmonary disease, or asthma; hematologic and oncologic disorders; pernicious anemia; clinically significant and unstable active gastrointestinal, renal, hepatic, endocrine, or cardiovascular system diseases; newly treated hypothyroidism;
* current or reported psychiatric (assessed by the SCID-II or neurological (assessed by a clinical neurological evaluation) disorders (e.g., schizophrenia, mood disorders, anxiety disorders, stroke, Parkinson's disease, seizure disorder, head injury with loss of consciousness, and any other significant mental or neurological disorder);
* known or suspected history of alcoholism or drug dependence and abuse during lifetime

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
functional Magnetic Resonance Imaging (fMRI) changes | at baseline, immediately after the intervention and after 3 days
  Changes in correlation of brain activity in different regions of brain as assessed by Blood Oxygenation Level Dependent (BOLD) signal.
  fMRI data are collected using gradient-echo echo-planar imaging at 3T (Philips Achieva) using a (T2*)-weighted imaging sequence sensitive to BOLD (TR = 3 s, TE = 30 ms, matrix = 80 x 80, FOV=224x224, slice thickness = 3 mm, flip angle = 90°, 50 slices, 240 vol).

SECONDARY OUTCOMES:
De-Blinding questionnaire | immediately after the intervention
  The questionnaire consists of three consecutive questions about subjects' perception of the treatment received. After being questioned on whether according to their perception, they thought they have received OMT or MP treatment, subjects were asked on a 0-10 numeric rating scale (NRS), where 0 represented absolutely uncertainty and 10 represented absolutely certainty, how certain they were regarding group allocation. Finally, they were asked to rate the perceived usefulness of the treatment received, based on a 0-10 NRS, where 0 represented absolutely useless and 10 represented absolutely useful

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Lucia Foundation I.R.C.C.S., Roma, Rm, Italy

IPD SHARING:
Plan to Share IPD: Undecided